CLINICAL TRIAL: NCT04747509
Title: Effects of Blackburn Exercises on Scapulothoracic Stability in Patients With Type-1 Scapular Dyskinesia
Brief Title: Blackburn Exercises in Type-1 Scapular Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00866 Rimsha Malik
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Scapular Dyskinesis
Keywords: Scapulothoracic stability; Blackburn exercises; Lateral scapular slide test; Type-1 Scapular Dyskinesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blackburn exercises (Experimental): Blackburn exercises and hot pack
  Interventions: Other: Blackburn exercises
- Conventional physical therapy (Active Comparator): Conventional physical therapy and hot pack
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: Blackburn exercises — Experimental group will include Blackburn exercises and hot pack for 10 minutes prior to the application of exercises; 3 sessions/week for a total of 4 weeks. Measurement will be taken at base level and after the last session, i.e. bilateral difference in lateral scapular slide test, serratus anterior and lower trapezius muscle strength, static measurements of scapula ROM, and pain and disability.
  These exercises will include prone horizontal abduction neutral and with full external rotation, prone horizontal scaption neutral and with full external rotation, prone horizontal external rotation, prone horizontal extension. All these exercises will be performed 3x15 repetitions with 30 seconds rest interval between each set.
  Arms: Blackburn exercises
Other: Conventional Physical therapy — Control group will include conventional physical therapy and hot pack for 10 minutes prior to the application of exercises; 3 sessions/week for a total of 4 weeks. Measurement will be taken at base level and after the last session, i.e. bilateral difference in lateral scapular slide test, serratus anterior and lower trapezius muscle strength, static measurements of scapula ROM, and pain and disability.
  These exercises will include push-ups on a stable surface, upward rotation shrugs and resisted scapular retraction. All these exercises will be performed 3x15 repetitions with 30 seconds rest interval between each set.
  Arms: Conventional physical therapy

SUMMARY:
The purpose of this study is to evaluate the effects of Blackburn exercises on Scapulothoracic stability in patients with Type-1 Scapular Dyskinesia, in comparison with conventional physical therapy. A randomized control trial is being conducted at National Institute of Rehabilitation Medicine (NIRM), Islamabad and Railway Hospital, Rawalpindi. The sample size was calculated through open epi tool, is 38. The participants are divided into two equal groups, 19 participants in experimental group and 19 participants in control group. The study duration is six months. Sampling technique applied is non-probability convenient sampling and groups have been randomized using sealed envelope method. Participants aged 25-55 years, having Type-1 Scapular Dyskinesia due to shoulder related causes, positive scapular assistance test, bilateral distance>1.5 cm in Lateral scapular slide test are being included in the study. Tools that are being used in this study are Lateral Scapular Slide Test, handheld dynamometer, Static measurements with scapula goniometry, and Shoulder pain and disability index (SPADI). Data will be analyzed through Statistical Package for Social Sciences (SPSS).

DETAILED DESCRIPTION:
The shoulder joint plays an important role in the function of the upper limb and in the activities of daily living. Shoulder pathologies are very common with the lifetime risk being between 40% and 60%. Prevalence rates of shoulder disorders are approximately 70% as compared to other musculoskeletal conditions. Ideal motion of scapula plays a major role in the shoulder functioning, any variation in the kinematics of scapula leads to various pathologies in shoulder and alteration in the scapular positioning can affect pain in the shoulder. Loss in the rhythmic functionality of the scapula due to muscular imbalance results in the scapular dyskinesia.

Scapular Dyskinesia is an observable alteration in the position of the scapula and the pattern of scapular motion in relation to the thoracic cage during static or dynamic movement of scapula. According to Borloz et al., a defective scapular posture caused by muscular imbalances, also generates imbalances of muscular strength. Scapular dyskinesia is followed by combination of symptoms such as malposition of scapula, prominent inferior border, pain in coracoids process and scapular motion dyskinesia. Patients report scapular medial border pain mainly. Kibler et al classified scapular dyskinesia in three dysfunctional patterns. Type I is characterized by posterior displacement or winging of the inferior medial scapular border. It is associated with inflexibility of pectoralis major and minor, and weakness of lower trapezius and serratus anterior. Type II is characterized by the projection of the entire medial border of the scapula. Type III is characterized by excessive superior translation, with elevation and some anterior displacement of the superior border of the scapula on the thorax. According to data reported in the literature, Scapular Dyskinesia (SD) incidence is frequent in patients with shoulder diseases, including rotator cuff diseases, glenohumeral instability, impingement syndrome, and labral tears. Type 1 pattern is however most commonly found in patients with rotator cuff dysfunction , shoulder impingement and instability, with the development of dyskinesis being associated with trapezius and serratus anterior, both of which are weakened in Type 1 Scapular Dyskinesia.

Generally the muscles that stabilize the scapula are directly related to direct-trauma, microtrauma, leading to muscle weakness and inhibition of movement by painful conditions around the shoulder. The serratus anterior and trapezius are the most susceptible to the effects of this inhibition, and are most often involved in the early stages of shoulder pathology. Stability at the scapulothoracic joint depends on the surrounding musculature. When the arm is raised overhead, the scapulothoracic motion involves upward rotation and posterior tilt of the scapula. Of the numerous muscles inserted on the scapula, those playing the most important role in the scapulothoracic kinematics are the upper and lower trapezius, and the serratus anterior. The serratus anterior (SA) works in concert with the upper and lower trapezius to upwardly rotate the scapula. Most overhead lifts and push-ups effectively recruit the serratus anterior. Activity of the serratus anterior tends to increase linearly with the amount of elevation at the glenohumeral joint. So when the scapulothoracic rhythm is altered, there are associated changes in glenohumeral angulation and loss of normal arm position, motion and stability.

In rehabilitation of scapular dyskinesia, therapeutic exercises should give attention to restoring the alignment of the scapulothoracic area and control of scapular muscles. The physiotherapy management is aimed to decrease the imbalances in the scapular stabilizing muscles so that control of scapular motion can be acquired. Interventions for scapular dyskinesia comprise of various stabilization exercises for scapula, but evidence scarcity is there in relation to Blackburn exercises in scapular dyskinesia. Blackburn exercises are one of the ways to treat shoulder pain and to regain proper mobility and decrease painful movements. These scapular stabilization exercises, based on stretching and strengthening, aim to improve muscle strength and joint position sense. The goal of increasing muscle strength is obtained with the aid of facilitation, and focus on restoring the alignment of the scapulothoracic area and control of scapular muscles. The Blackburn exercises are optimal for the stimulation of lower trapezius, being the "Y" the optimal exercise for this purpose. However, there is no clear evidence regarding their effect on serratus anterior. Although serratus anterior muscle works in concert with lower trapezius, and it is the only scapulothoracic muscle that produces upward rotation of the scapula with acromioclavicular (AC) joint external rotation and posterior tilting.

There is dearth in literature regarding the effect of Blackburn exercises on scapulothoracic stability in Dyskinesia, in relation to serratus anterior and lower trapezius muscles. There is poor available evidence regarding the effects of Blackburn exercises specifically on serratus anterior muscle strength, contributing to scapulothoracic stability. Also, the studies conducted previously were lacking a control group for comparison, and majority of the intervention protocols evaluated the immediate effects of Blackburn exercises with no focus on scapular stabilizers.

Literature Review:

A case report presented by Navreet Kaur et al. in 2019 evaluated the effects of Blackburn exercises in scapular dyskinesia. By the end of one week of treatment, the patient felt no pain in resisted movements and range of motion was complete. After one month of treatment, observations included both shoulders on the same level, no droop observed from antero-posterior view and no prominency of scapular border from postero-anterior view.

In 2018, Rasika Panse et al evaluated the effects of Blackburn exercises in shoulder impingement in rock climbers on pain and disability using Shoulder pain and disability index (SPADI) scale. Subjects were given Blackburn exercises thrice a week with each session lasting for 30 minutes. They reported positive results of Blackburn exercises in shoulder impingement, with decreased pain in certain shoulder movements after treatment. However, long term effects and the effects of Blackburn exercises on shoulder muscles were not considered.

Another study was conducted by Patel Neelam Jayesh et al. regarding the effectiveness of open kinematic chain exercises in overhead atheletes with SICK scapula. Participants were given 4 sessions per week for 3 weeks and the intervention protocol included Blackburn exercises along with Dynamic hug, W exercise, Lunges with dumbells and Pectoralis minor stretching. Results of this study showed significant improvement after 3 weeks of intervention.

Pradeep Shankar et al conducted a study to find the effect of scapular stabilization exercises for Type 2 Scapular Dyskinesia in subjects with shoulder impingement. 3 sessions of scapular stabilization exercises were given per week for 2 weeks and outcomes were measured using Lateral Scapular Slide Test and Shoulder pain and disability index (SPADI). Study findings reported the protocol to be effective. However this study lacked a control group receiving only conventional exercises. Also, the study was done for a period of two weeks, therefore long term effects were not known.

In 2018, Hugo Machado Sanchez reviewed the Scapular Dyskinesia from the point of view of pathology, evaluation and treatment. He concluded that emphasis on strengthening of scapular depressor muscles and scapular stabilizers acting primarily on the shoulder should be of paramount importance for the restoration of normal scapular function in rehabilitation of Scapular Dyskinesia.

Kevin G. Laudner et al. assessed the relationship between lower trapezius and serratus anterior strength and the quantity of scapular upward rotation by using a hand-held dynamometer. The results of their study demonstrated a moderate-good relationship between scapular upward rotation and lower trapezius strength. However, a poor relationship was seen between scapular upward rotation and serratus anterior strength that was thought to be due to strength measurement occurring at a higher amount of humeral elevation (120°-130°) than was tested during scapular upward rotation (0° , 60° , 90° , 120°).

ELIGIBILITY:
Inclusion Criteria:

* Type-1 Scapular Dyskinesia patients with shoulder related causes
* Positive scapular assistance test
* Bilateral difference > 1.5 cm in Lateral Scapular Slide Test

Exclusion Criteria:

* Non-shoulder related scapular dyskinesia
* Recent fracture or trauma
* Malignancy
* Severe systemic illness
* Corticosteroid injections in the affected shoulder in the preceding 6-9 weeks
* Any other medically diagnoses orthopaedic, neurological or cardiovascular disorder affecting upper extremity function

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Lateral Scapular Slide Test | 12th day
  Changes from baseline bilateral scapular distance are taken with the help of tape measure.
Handheld Dynamometer | 12th day
  Changes from baseline grip strength are taken with the help of hand dynamometer.
Static Measurements with Scapular Goniometry | 12th day
  Changes from baseline measurements of infera, lateral displacement and abduction are taken with the help of tape measure and goniometer.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 12th day
  It was developed to measure current shoulder pain and disability in an outpatient setting. It consists of a 5-item subscale that measures pain and an 8-item subscale that measures disability. Pain scale is summed up to a total of 40 and disability scale to 80. A total score of 0 indicates best and 100 indicates worst.

OTHER OUTCOMES:
Manual Muscle Testing | 12th day
  Changes from the baseline serratus anterior and lower trapezius are taken according to manual muscle testing grading system. Grading Scale Range: 0 to 5 0: None: No visible or palpable contraction,
  1. Trace: Visible or palpable contraction with no motion
  2. Poor: Full ROM gravity eliminated
  3. Fair: Full ROM against gravity
  4. Good: Full ROM against gravity, moderate resistance
  5. Normal: Full ROM against gravity, maximul resistance

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PHD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - National Institute of Rehabilitation Medicine (NIRM), Islamabad, Federal
  - Railway General Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panagiotopoulos AC, Crowther IM. Scapular Dyskinesia, the forgotten culprit of shoulder pain and how to rehabilitate. SICOT J. 2019;5:29. doi: 10.1051/sicotj/2019029. Epub 2019 Aug 20. PMID 31430250
- [Background] Kaur N. Effect of Blackburn Exercises in Scapular Dyskinesia: a case report. Journal of the Gujarat Research Society. 2019 Dec 24;21(8):961-7.
- [Background] Borloz S, Graf V, Gard S, Ziltener JL. [Scapular dyskinesis]. Rev Med Suisse. 2012 Dec 19;8(367):2422-8. French. PMID 23346745
- [Background] Shankar P, Jayaprakasan P, Devi R. Effect of scapular stabilisation exercises for type 2 scapular dyskinesis in subjects with shoulder impingement. International Journal of Physiotherapy. 2016 Feb 1;3(1):106-10.
- [Background] Longo UG, Risi Ambrogioni L, Berton A, Candela V, Massaroni C, Carnevale A, Stelitano G, Schena E, Nazarian A, DeAngelis J, Denaro V. Erratum: Longo, U.G., et al. Scapular Dyskinesis: From Basic Science to Ultimate Treatment. International Journal of Environmental Research and Public Health 2020, 17(8), 2974. Int J Environ Res Public Health. 2020 May 27;17(11):3810. doi: 10.3390/ijerph17113810. PMID 32471164
- [Background] Sanchez HM, Sanchez EG. Scapular dyskinesis: biomechanics, evaluation and treatment. Int Phys Med Rehab J. 2018;3(6):514-20.
- [Background] Jayesh PN, Muragod AR, Motimath B. Open kinematic chain exercises for SICK scapula in competitive asymptomatic over head athletes for 3 weeks. Int J Physiother Res. 2014;2(4):608-15.
- [Background] Postacchini R, Carbone S. Scapular dyskinesis: diagnosis and treatment. OA Musculoskeletal Medicine. 2013 Oct 18;1(2):20.
- [Background] Manske RC, Grant-Nierman M, Lucas B. Shoulder posterior internal impingement in the overhead athlete. Int J Sports Phys Ther. 2013 Apr;8(2):194-204. PMID 23593557
- [Background] Panse R, Yeole U, Pawar K, Pawar P. Effects of Blackburn exercises in shoulder impingement on pain and disability in rock climbers. Age. 2018;22:3-57.
- [Background] Laudner KG, Stanek JM, Meister K. The relationship of periscapular strength on scapular upward rotation in professional baseball pitchers. J Sport Rehabil. 2008 May;17(2):95-105. doi: 10.1123/jsr.17.2.95. PMID 18515910